CLINICAL TRIAL: NCT05757921
Title: Non-surgical Treatment of Periodontitis With or Without the Adjunctive Treatment of Perisolv®
Brief Title: Comparison of Adjunctive Chemomechanical Therapy With Standard Care in Patients With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristianstad University (Other)
Responsible Party: Principal Investigator, Viveca Wallin Bengtsson, Principle investigator, Kristianstad University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Peri_Solv
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Periodontitis
Keywords: probing pocket depth; bleeding on probing; dental plaque
MeSH Terms: conditions — Periodontitis; Dental Plaque

STUDY DESIGN:
Intervention Model Description: Test group: non-surgical mechanical treatment and adjunctive treatment Perisolv Control group: non-surgical mechanical treatment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Principal investigator and investigator (the periodontologists) were calibrated prior to the study.
  Outcome assessments were performed separately by the periodontologists and blinded. The statisticians were also blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-surgical mechanical treatment with Perisolv® (A) (Experimental): The test group will receive the following treatment: In the deepened pockets to be treated, Perisolv is initially applied according to the manufacturers recommendation.Then subgingival debridement is performed. This is performed with piezoelectric ultrasound (EMS) while rinsing water and completed with subgingival manual instrumentation. In addition an aliquot of Perisolv was left after final debridement.
  Interventions: Device: Perisolv (A)
- Non-surgical mechanical treatment without Perisolv® (B) (Active Comparator): The control group will receive the following treatment: In the deepened pockets to be treated, subgingival debridement is performed. This is performed with piezoelectric ultrasound (EMS) while rinsing water and completed with subgingival manual instrumentation.
  Interventions: Other: Standard (B)

INTERVENTIONS:
Device: Perisolv (A) — Intended for cleaning periodontal pockets for both periodontitis and peri-implantitis. Softens degenerative tissue and biofilm before depuration of periodontal pockets. Does not affect healthy tissue.
  Arms: Non-surgical mechanical treatment with Perisolv® (A)
Other: Standard (B) — Deepened periodontal pockets to be treated are performed by subgingivally debridement. This is performed with piezoelectric ultrasound (EMS) under rinsing water and subgingival debridement with hand instrument.
  Arms: Non-surgical mechanical treatment without Perisolv® (B)

SUMMARY:
The goal of the clinical trial is to compare adjunctive chemomechanical therapy with standard care regarding root planning in patients with periodontitis. The primary outcome is to measure pocket depth before and after treatment in the test, and control group respectively

Secondary outcomes:

* Bleeding on probing
* Plaque index
* Quality of life from standardized protocol

The hypothesis is that non- surgical mechanical treatment with chloramines in patients with periodontitis will show a better pocket closure after the treatment.

DETAILED DESCRIPTION:
Data from the clinical treatment were registered in patient records. In parallel, clinical data were documented in a study protocol and saved in a safe in accordance with standard operation procedure at the clinic.The protocol with medical records were not opened until the study was completed and only by authorized persons with access to the data in the study such as, principal investigator and statisticians.

Variables used in the study originates from an international working group in periodontology in 2018 (Papapanou PN, et al 2018). In accordance with the working group diagnosis of periodontitis should include pocket depth, bleeding, and bone loss (X-ray). Thus, in this study the primary outcomes were pocket depth and bleeding on probing.

To compare scaling and root planning in periodontitis with an adjunctive application to enhance the standard care; an active comparator (Control group) was compared with an experimental arm (Test group).

Patients were therefore randomized into a test or control group. Inclusion criteria

* At least four pathological pockets ≥ 5 mm and bleeding on probing Exclusion criteria
* Diabetes HbA1c >7.0, antibiotics 3 months before treatment, cortisone treatment and if needed prophylactic antibiotics

Patients that participated in the study were consecutively given an ID code. Data was collected and registered in the ordinary patient journal. Journal entry and a research protocol was used with the unique ID number as to prevent breaches of privacy. The dental hygienist performed the treatments and was therfore not blinded. The periodontologists performed the primary and secondary outcomes within the clinical study were both blinded. The code list with the actual treatment was secured in a locked up space, at the clinic. Upon the final appointment the specific arm of treatment was registered by the dental hygienist in the patient journal. To ensure that the data from the study were correctly registered three independent dental nurses were validating the data separately.

All patients were given oral and written information about the study and signed a written informed consent. The patients were informed that they could drop off whenever they wanted without any explanations. The ethical board approved the study.

From a standard operation procedure by good clinical practice and Swedish legislation (The national board of social affairs and health and Health and Medical Care Act), the control group was exposed to mechanical non-surgical treatment in addition with oral hygiene instructions at baseline, 3 months, and 12 months. In the test group the same standard operation procedure was performed with the addition of Perisolv® in all pathological pockets ≥ 4 mm. Perisolv® was added initially and directly after the treatment. At all-time points both primary and secondary outcomes were determined for all pockets. In addition, the instrument Oral Health Impact Profile (OHIP) was used as a measurement of quality of life.

Risk assessments was handled by the safety regulation and quality plan of the clinic.The clinic followed the Swedish legalisation, Health and Medical Care Act with quality assurance. If any adverse events during the treatments the local standard operation procedures ensured reporting to concerned authority in Sweden. Participant not fulfilling the study was reported in the patient journal as not completed and statistically noted as missing data.

Regarding the study's safety plan any adverse event during the treatment code list would be decoded and would be covered by the dental insurance.

From the power analysis 32 individuals were minimum to reach a clinically significant difference at 0.5 mm between the groups with alpha 0.05 and power 80%. The IBM SPSS version 27.0 statistical software package (SPSS Inc., Armonk, NY, USA) for personal computer was used in the statistical analyses. Statistics was calculated as means with standard deviation (SD). Independent t-tests (equal variance not assumed) paired t-test and one-way ANOVA test were used to compare inter and intra-group differences. Non-parametric chi-square test was used for categorical variables. Statistical significance was set with 80 percent at p < 0.05. Non visits were recorded as missing data in the statistics.

ELIGIBILITY:
Inclusion Criteria:

Individuals who agree to participate in the study and who also have at least 4 gingival pockets with probing depth ≥5 mm and which at the same time bleed on probing.

-

Exclusion Criteria:

* Individuals with uncontrolled/difficult diabetes mellitus (HbA1c > 7.0)
* Individuals who need antibiotic prophylaxis
* Individuals taking medication with Prednisolone.
* Individuals taking medication that has a known side effect, gingival hyperplasia
* Individuals who took systemic antibiotics 3 months before the start of the study.

Min Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-10-24 (Actual); Primary Completion 2014-05-16 (Actual); Study Completion 2014-05-16 (Actual)

PRIMARY OUTCOMES:
probing pocket depth | baseline
  millimeter
probing pocket depth | 3 months
  millimeter
probing pocket depth | 12 months
  millimeter

SECONDARY OUTCOMES:
bleeding on probing | baseline
  percent
bleeding on probing | 3 months
  percent
bleeding on probing | 12 months
  percent
plaque index | baseline
  percent
plaque index | 3 months
  percent
plaque index | 12 months
  percent

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Marie AJ Roos Jansaker, Assoc.Prof., Principal Investigator — Kristianstad University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smiley CJ, Tracy SL, Abt E, Michalowicz BS, John MT, Gunsolley J, Cobb CM, Rossmann J, Harrel SK, Forrest JL, Hujoel PP, Noraian KW, Greenwell H, Frantsve-Hawley J, Estrich C, Hanson N. Systematic review and meta-analysis on the nonsurgical treatment of chronic periodontitis by means of scaling and root planing with or without adjuncts. J Am Dent Assoc. 2015 Jul;146(7):508-24.e5. doi: 10.1016/j.adaj.2015.01.028. PMID 26113099
- [Background] Ferreira MC, Dias-Pereira AC, Branco-de-Almeida LS, Martins CC, Paiva SM. Impact of periodontal disease on quality of life: a systematic review. J Periodontal Res. 2017 Aug;52(4):651-665. doi: 10.1111/jre.12436. Epub 2017 Feb 8. PMID 28177120
- [Background] Citterio F, Gualini G, Chang M, Piccoli GM, Giraudi M, Manavella V, Baima G, Mariani GM, Romano F, Aimetti M. Pocket closure and residual pockets after non-surgical periodontal therapy: A systematic review and meta-analysis. J Clin Periodontol. 2022 Jan;49(1):2-14. doi: 10.1111/jcpe.13547. Epub 2021 Nov 11. PMID 34517433
- [Background] Jepsen K, Jepsen S. Antibiotics/antimicrobials: systemic and local administration in the therapy of mild to moderately advanced periodontitis. Periodontol 2000. 2016 Jun;71(1):82-112. doi: 10.1111/prd.12121. PMID 27045432
- [Background] Guida A. Mechanism of action of sodium hypochlorite and its effects on dentin. Minerva Stomatol. 2006 Sep;55(9):471-82. English, Italian. PMID 17146426
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Derived] Wallin-Bengtsson V, Scherdin-Almhojd U, Roos-Jansaker AM. Supra- and sub-gingival instrumentation of periodontitis with the adjunctive treatment of a chloramine - a one-year randomized clinical trial study. Acta Odontol Scand. 2024 Mar 22;83:1-6. doi: 10.1080/00016357.2023.2281486. PMID 37962876